CLINICAL TRIAL: NCT03297996
Title: The Gut Microbiota in Conventional and Serrated Precursors of Colorectal Cancer
Brief Title: Study of Gut Microbiome and Colorectal Tumors
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 11-01377
Record Dates: First submitted 2017-09-27; First posted 2017-09-29 (Actual); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Serrated Polyp; Hyperplastic Polyp; Sessile Serrated Adenoma; Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA was extracted from stool using the PowerLyzer PowerSoil Kit (Mo Bio Laboratory Inc., CA) following the manufacturer's protocol. DNA was collected and eluted using silica columns included with the PowerLyzer PowerSoil kit. Barcoded amplicons were generated covering the V4 region of the 16S rRNA gene using the F515/R806 primer pair.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SIT: Centers for Disease Control and Prevention (CDC) Study of In-home Tests for Colorectal Cancer (SIT)
  Interventions: Diagnostic Test: Mobio PowerSoil DNA Isolation Kit
- NYU: New York University (NYU) Human Microbiome and Colorectal Tumor study
  Interventions: Diagnostic Test: Mobio PowerSoil DNA Isolation Kit

INTERVENTIONS:
Diagnostic Test: Mobio PowerSoil DNA Isolation Kit — 16S rRNA amplicons covering variable regions V3 to V4 were generated using primers (347F-5'GGAGGCAGCAGTRRGGAAT'-3' and 803R 5'-CTACCRGGGTATCTAATCC-3') incorporating Roche 454 FLX Titanium adapters (Branford, CT) and a sample barcode sequence

SUMMARY:
Gut microbiota were assessed in 540 colonoscopy-screened adults by 16S rRNA gene sequencing of stool samples. Investigators compared gut microbiota diversity, overall composition, and normalized taxon abundance among these groups.

DETAILED DESCRIPTION:
Colorectal cancer is a heterogeneous disease arising from at least two precursors-the conventional adenoma (CA) and the serrated polyp. A relationship between the human gut microbiota and colorectal cancer has been shown; however, its relationship to the different early precursors of colorectal cancer is understudied. This study tested, for the first time, the relationship of the gut microbiota to specific colorectal polyp types.

ELIGIBILITY:
Inclusion Criteria:

* Both men and women who have visited a gastroenterologist or surgeon, aged 18 or older will be included in this study.
* Both men and women residents in the United States, aged 18 or older will be included in this study.

Exclusion Criteria:

* Women who are pregnant will be excluded from participating in this study
* Subjects on ongoing antibiotic therapy will be excluded from participating in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: There are no enrollment restrictions based on race or ethnic origins. Vulnerable subjects such as pregnant women and children will not be involved in this study. We will not ask subjects about sensitive topics such as Mental Health, drug/alcohol abuse, or others that fall in this category.
Sampling Method: Non-Probability Sample
Enrollment: 540 (Actual)
Dates: Start 2011-11-23 (Actual); Primary Completion 2015-04-25 (Actual); Study Completion 2015-04-25 (Actual)

PRIMARY OUTCOMES:
Prevalence and relative abundance of selected fecal microbial taxa | 2 Days
  Quantitative polymerase chain reaction

CONTACTS AND LOCATIONS:
Overall Officials: Jiyoung Ahn, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States